CLINICAL TRIAL: NCT05270070
Title: A Pilot Study: Comparing Digital to Traditional Booking System for Clinical Appointments
Brief Title: Digital Versus Traditional Booking System for Clinical Appointments
Status: Completed | Type: Observational
Sponsor: Canadian Forces Health Services Centre Ottawa (Other)
Collaborators: Canadian Department of National Defence (Other Government)
Responsible Party: Principal Investigator, Gaurav Gupta, Principal Investigator, Canadian Forces Health Services Centre Ottawa
Other Study IDs: E2021-11-048-008-0002
Record Dates: First submitted 2022-02-11; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Health Informatics
Keywords: digital booking; telephone booking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Digital Booking: Patients bookings done through digital booking system.
  Interventions: Other: Appointment booking system
- Traditional Booking: Patients bookings done through traditional booking like telephone or secure email.
  Interventions: Other: Appointment booking system

INTERVENTIONS:
Other: Appointment booking system — Patients were sent an email to book an appointment using the telephone/email versus a online booking system.

SUMMARY:
In the Canadian Forces Health Services Ottawa clinical administrative resources are currently constrained, directly impacting workflow and patient care. Given the nature of the current EMR and digital health infrastructure, DBS is not currently being employed. Therefore, investigators sought to determine the relative benefit of using an online booking system when compared to TB. To the investigator's knowledge, validation of this type has not been conducted in this setting.

DETAILED DESCRIPTION:
Introduction: The impact of digital booking systems (DBS) on clinical care, administrative efficiency and health care costs have not previously been explored in the Canadian Forces Health Services. No show rates were shown to be reduced by 6-42% percent compared to traditional booking (TB) depending on the system and the clinic. Therefore, investigators sought to determine the relative benefit of using an online booking system when compared to TB.

Methods: Main outcome variables included total time for booking all patients between groups including the start to end dates of each intervention, the number of hours spent on the phone / answering emails, and the number of phone calls and emails received, and the number of phone calls / emails regarding booking problems, cancellations, changes and no shows. Descriptive and mean comparative statistics will be used to determine any differences between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have never been seen for new consultations

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred to the Canadian Forces Health Services Centre for physical medicine and rehabilitation consultation.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Total time for booking all patients | ~3 months
  total time taken for DB and TB patients to be booked in a clinic time slot

SECONDARY OUTCOMES:
Percent of Patients Booked | ~3 months
  Percent of Patients Booked for each group
Average Time Spent per Patient | ~3 months
  Average Time Spent per Patient

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Gupta, MD, Principal Investigator — Canadian Forces Health Services Centre
Locations (1):
- Canadian Forces Health Services Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No